CLINICAL TRIAL: NCT07344974
Title: A Randomized Controlled Single-Center Clinical Trial of Traditional Chinese Medicine Hand and Foot Bath for Taxane-Induced Peripheral Neurotoxicity
Brief Title: Hand and Foot Bath for Taxane-Induced Peripheral Neurotoxicity
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025YJZ98
Record Dates: First submitted 2025-11-19; First posted 2026-01-15 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; Chemotherapy-induced peripheral neuropathy; Traditional Chinese Medicine
MeSH Terms: conditions — Breast Neoplasms | interventions — Medicine, Chinese Traditional; mecobalamin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TCM arm (Experimental)
  Interventions: Drug: Traditional Chinese medicine (TCM) hand and foot baths
- methylcobalamin arm (Active Comparator)
  Interventions: Drug: Methylcobalamin (methylB12)

INTERVENTIONS:
Drug: Traditional Chinese medicine (TCM) hand and foot baths — Traditional Chinese medicine (TCM) formula "Yi-Qi Yang-Xue Tong-Luo Fang" hand and foot baths
  Arms: TCM arm
Drug: Methylcobalamin (methylB12) — methylcobalamin is a commonly used neurotrophic agent in CIPN
  Arms: methylcobalamin arm

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common and dose-limiting toxicity of taxane-based agents, with an incidence of 57%-83%. Patients frequently develop fingertip numbness, reduced tactile sensation, and other neuropathic symptoms, which significantly impair quality of life. The severity of CIPN is strongly associated with cumulative drug dosage. Current management strategies remain inadequate, and no high-level clinical recommendations are available.

Traditional Chinese medicine (TCM) hand and foot baths have been widely applied in clinical practice due to their convenience, low cost, and high patient acceptance. The formula "Yi-Qi Yang-Xue Tong-Luo Fang," developed by the TCM Department of our hospital. Preliminary clinical use has shown reliable efficacy and good tolerability, suggesting potential benefit for CIPN.

This randomized, controlled clinical trial aims to evaluate the efficacy and safety of the TCM hand and foot bath compared with methylcobalamin (a commonly used neurotrophic agent) for paclitaxel-induced CIPN. Peripheral neurotoxicity will be assessed using standardized measures, including the Common Terminology Criteria for Adverse Events (CTCAE), the Total Neuropathy Score-clinical version (TNSc), and the M. D. Anderson Symptom Inventory with TCM module (MDASI-TCM). Changes in scores between groups will be compared to determine relative effectiveness.

Quality of life will be evaluated using validated international scales, specifically the EORTC Quality of Life Questionnaire for Breast Cancer Patients (EORTC QLQ-BR23) and the core questionnaire (EORTC QLQ-C30). These tools will provide multidimensional evaluation of treatment impact on daily functioning and well-being.

The study is expected to generate evidence on both efficacy and safety of this TCM formula, clarify its potential role in preventing or reducing CIPN progression, and assess its influence on patients' quality of life. The findings will provide clinical data to support TCM-based interventions as complementary strategies for managing chemotherapy-induced neurotoxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed breast cancer;
2. Development of grade ≥1 peripheral neurotoxicity after receiving a taxane-containing regimen, with continuation of this regimen for at least two additional cycles;
3. Age ≥18 years, male or female;
4. ECOG performance status score 0-1;
5. Adequate major organ function (cardiac, hepatic, renal, and bone marrow) within 7 days before treatment, meeting the following requirements:

   1. Hematology (without blood transfusion within the previous 14 days):
   2. Hemoglobin (Hb) ≥90 g/L;
   3. Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L;
   4. Platelets (PLT) ≥75 × 10⁹/L.
6. Biochemical tests:

   1. Total bilirubin (TBIL) ≤1.5 × upper limit of normal (ULN);
   2. ALT and AST ≤2.5 × ULN;
   3. Serum creatinine (Cr) ≤1.5 × ULN or creatinine clearance (CCr) ≥60 mL/min.
7. Estimated survival ≥6 months;
8. Signed informed consent.

Exclusion Criteria:

1. Pre-existing neurological disorders, including peripheral or central neuropathy;
2. Known allergy to components of the investigational TCM formula;
3. Neuropathy caused by electrolyte imbalance, diabetes, or other metabolic diseases;
4. Neuropathy due to nerve compression of any cause;
5. Concomitant use of other neuroprotective therapies (e.g., nerve growth factor, vitamin B, calcium-magnesium preparations);
6. Pregnant or lactating women;
7. Cognitive impairment or psychiatric disorders;
8. Any other condition considered unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With Controlled Peripheral Neurotoxicity at Week 6 as Assessed by CTCAE v5.0 | From baseline (within 7 days before the first administration of study drug) to 6 weeks ±7 days after treatment initiation; assessments will continue every 6 weeks until 6 weeks after the last cycle of taxane chemotherapy.
  Peripheral neurotoxicity will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Neurotoxicity progression is defined as an increase of ≥1 CTCAE grade from baseline. Controlled peripheral neurotoxicity is defined as stable or improved CTCAE grade compared with baseline. The outcome will be summarized as the proportion of participants with controlled peripheral neurotoxicity at week 6.
Proportion of Participants With Controlled Peripheral Neurotoxicity at Week 6 Assessed by the MD Anderson Symptom Inventory-Traditional Chinese Medicine Module (MDASI-TCM) | From baseline (within 7 days before the first administration of study drug) to 6 weeks ±7 days after treatment initiation; assessments will continue every 6 weeks until 6 weeks after the last cycle of taxane chemotherapy.
  Symptom severity will be assessed using the MD Anderson Symptom Inventory-Traditional Chinese Medicine module (MDASI-TCM). Changes in symptom burden will be evaluated by comparing MDASI-TCM scores from baseline to week 6. The outcome will be summarized as the proportion of participants with controlled peripheral neurotoxicity in MDASI-TCM score at week 6.
Proportion of Participants With Controlled Peripheral Neurotoxicity at Week 6 as Assessed by Total Neuropathy Score-Clinical Version (TNSc) | From baseline (within 7 days before the first administration of study drug) to 6 weeks ±7 days after treatment initiation; assessments will continue every 6 weeks until 6 weeks after the last cycle of taxane chemotherapy.
  Peripheral neuropathy severity will be assessed using the Total Neuropathy Score-Clinical version (TNSc). Changes in peripheral neuropathy severity will be evaluated by comparing TNSc scores from baseline to week 6. The outcome will be summarized as the proportion of participants with controlled peripheral neurotoxicity at week 6.

SECONDARY OUTCOMES:
Time to Peripheral Neurotoxicity Progression as Assessed by CTCAE v5.0 | From the first administration of study drug to the date of first documented neurotoxicity progression, as assessed by CTCAE criteria, up to 6 weeks after the last cycle of taxane chemotherapy.
  Time to peripheral neurotoxicity progression is defined as the time interval from the first administration of the study intervention to the first documented occurrence of peripheral neurotoxicity progression, as assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Neurotoxicity progression is defined as an increase of ≥1 CTCAE grade from baseline. Participants without documented progression will be censored at the date of the last neurotoxicity assessment.
Change from Baseline in Quality of Life Scores (EORTC QLQ-C30 and QLQ-BR23) | From baseline (within 7 days before treatment initiation) to every 2 chemotherapy cycles, until 6 weeks after the last taxane chemotherapy.
  Quality of life will be assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) and the Breast Cancer-Specific Module (EORTC QLQ-BR23).
  Changes in global health status and functional and symptom scales from baseline will be analyzed to evaluate the impact of the intervention on patients' quality of life.
Incidence of Adverse Events | From the first administration of study drug to 6 weeks after the last taxane chemotherapy cycle.
  All adverse events (AEs) occurring during the study will be recorded, including onset date, duration, severity (graded per CTCAE v5.0), management, and outcome. Investigators will assess the causal relationship between each AE and the study treatment, and document all findings in the case report form with signature and date.
  The number and percentage of participants experiencing treatment-related AEs will be summarized by severity grade and system organ class.